CLINICAL TRIAL: NCT05331586
Title: Remotely Monitored and Exercise Program in Gestational Weight Gain in Pregnant Women With Obesity
Brief Title: Remotely Monitored Exercise Program in Pregnant Women With Obesity
Acronym: GROB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0000
Record Dates: First submitted 2022-03-03; First posted 2022-04-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy Related; Obesity, Maternal
Keywords: Obesity; pregnancy; exercise; physical activity; maternal; gestational weight gain; gestational diabetes mellitus
MeSH Terms: conditions — Pregnancy in Obesity; Obesity; Motor Activity; Gestational Weight Gain; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control intervention (No Intervention): The control group will receive the standard prenatal care in Hospital Center of São Joao (CHUSJ). The standard prenatal care will be regular appointments with obstetrician and midwife nurses, ultrasounds and nutritional appointments. The pregnant women in control group will also receive a pamphlet with the benefits of physical exercise during pregnancy and recommendations for adequate gestational weight gain. Pregnant women in control group will not be discouraged from exercising on their own.
- Exercise intervention (Experimental): The exercise group intervention will perform home-based remotely monitored exercise
  Interventions: Behavioral: Remote Exercise

INTERVENTIONS:
Behavioral: Remote Exercise — The pregnant women will perform a home-based structured exercise programme. The exercise will be remotely monitored since the first gestational trimester until delivery
  Arms: Exercise intervention

SUMMARY:
Pregnant women with obesity will be invited to participate in structured home-based exercise programme, remotely monitored

DETAILED DESCRIPTION:
Pregnant women with obesity will be invited to participate in structured home-based exercise programme, remotely monitored. The remote system use inertial motion trackers, digitizes pregnant women motion and provides real-time feedback on performance through a mobile app. It also includes a web-based platform that allows the clinical team to prescribe, monitor and adapt the exercise program remotely. This way, the system allows patients to perform independent exercise program at home without the need for constant therapist supervision, ensuring remote monitoring throughout the rehabilitation program. The exercise programme will be performed since the first gestational trimester until delivery.

Data of gestational weight gain, gestational diabetes mellitus, low back pain and quality of life will be colected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with obesity (BMI ≥ 30 kg/m2) at first gestational trimester

Exclusion Criteria:

* pre-pregnancy BMI < 30 kg/m2;
* previous bariatric surgery;
* hemodynamically significant heart disease;
* restrictive lung disease;
* incompetent cervix or cerclage;
* multiple gestation;
* persistent second- or third-trimester bleeding;
* placenta previa after 26 weeks of gestation;
* premature labor during the current pregnancy;
* ruptured membranes;
* preeclampsia or pregnancy-induced hypertension;
* severe anemia;
* inability to read and understand Portuguese; ->15 weeks gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Gestational Weight Gain | At delivery
  Using portable digital scale (Tantita InnerScan BC-545). Gestational weight gain will be calculated as the difference between maternal weight at last appointment (36-39 gestational weeks) and pre-pregnancy weight.
Excessive gestational weight gain | At delivery
  The adequate gestational weight gain in pregnant women with obesity should not exceed 9kg in entire pregnancy, the values over these thresholds will be considered excessive gestational weight gain.

SECONDARY OUTCOMES:
Low Back Pain | At first, second and third gestational trimester
  Oswestry Low Back Pain Disability Questionnaire (ODI v2.0)
Subjective Physical Activity assessment | At first, second and third gestational trimester
  Pregnancy Physical Activity Questionnaire (PPAQ) is a self-reported questionnaire. The objective is measure the type and intensity of pregnant women physical activity.
Objective Physical Activity assessment | At first, second and third gestational trimester
  Accelerometry, is a device that monitors the acceleration of body segments, it is considered the gold standard with regard to objectivity and reliability (ICC:0.661-0.806)
Gestational Diabetes Mellitus | Second gestational trimester
  The presence of gestational diabetes mellitus will be assessed between 24-28 gestation weeks, through the Oral Glucose Tolerance Test. Blood sampling for fasting glucose concentrations will be taken after a 10 hour overnight fast, and glucose tolerance will measured by a 2 hours 75 mg per-oral glucose tolerance test. GDM will be diagnosed as fasting glucose ≥ 126 mg/dl or 2h concentration ≥ 200 mg/dl.
Quality of Life Assessment | At first, second and third gestational trimester
  COOP-Quality of life during Pregnancy Questionnaire
Pelvic Floor and sexual disorders during pregnancy | At first, second and third gestational trimester
  Assessment of Pelvic Floor Disorders and Their Risk Factors During Pregnancy and Postpartum Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Diana Bernardo, Porto, Portugal